CLINICAL TRIAL: NCT06483204
Title: Steroids for Rhinoplasty: Pain, Nausea, Edema and Ecchymosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was never started
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Priyesh Patel, Dr. Priyesh N. Patel, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #240474
Record Dates: First submitted 2024-06-25; First posted 2024-07-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Edema; Bruising; Nasal Obstruction; Postoperative Pain; Postoperative Nausea; Postoperative Complications
MeSH Terms: conditions — Edema; Contusions; Nasal Obstruction; Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Complications | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Medrol dosepak group (Experimental): For the experimental group, they will be given a medrol dosepak which is a prescription of oral steroids taken over a week long period. The dosage of steroids decreases each day. They will also complete a study survey each day remarking on our outcomes of interest such as facial swelling, bruising, pain, and nausea.
  Interventions: Drug: Medrol 4 MG Oral Tablet Includes Medrol Dosepak
- No medrol dosepak group (No Intervention): This group will not receive the medrol dosepak. They will still complete the daily survey until they return for their postoperative appointment, one week after their surgery.

INTERVENTIONS:
Drug: Medrol 4 MG Oral Tablet Includes Medrol Dosepak — Medrol tapered dosepak given to experimental arm patients to determine if there is a significant difference in pain, nausea, edema and ecchymosis outcomes in the postoperative period after a functional rhinoplasty procedure.
  Other Names: methylprednisolone
  Arms: Medrol dosepak group

SUMMARY:
This study will be a prospective randomized study to evaluate the effect of medrol dosepaks (oral corticosteroids) on postoperative outcomes among patients undergoing rhinoplasty by Facial Plastic Surgeons at Vanderbilt. Outcomes will include postoperative pain, nausea, and patient experience, with secondary outcomes of swelling and bruising.

Methylprednisolone is an oral corticosteroid that has been shown in multiple RCTs and is used extensively that it can significantly reduce postoperative swelling and bruising in postoperative rhinoplasty patients, however, we have not examined if those effects extend to their pain ratings, nausea, and overall patient experience. Current research on use of steroids in rhinoplasty suggests that its use may decrease pain and nausea and benefit the patients overall experience.

Minimizing complications for any surgery is of upmost importance for surgeons.. However, the benefits of oral corticosteroid use for rhinoplasty patients in the immediate post-operative period are poorly understood and practice patterns vary widely. To identify and quantify the benefits and drawbacks of oral corticosteroid use in the immediate post-operative period for primary rhinoplasty patients, pain, swelling, nausea, patient experience, and post-operative swelling will be studied.

DETAILED DESCRIPTION:
This study will be a prospective randomized study to evaluate the effect of medrol dosepaks (oral corticosteroids) on postoperative outcomes among patients undergoing rhinoplasty by Facial Plastic Surgeons at Vanderbilt. Outcomes will include postoperative pain, nausea, and patient experience, with secondary outcomes of swelling and bruising.

Methylprednisolone is an oral corticosteroid that has been shown in multiple RCTs and is used extensively that it can significantly reduce postoperative swelling and bruising in postoperative rhinoplasty patients, however, we have not examined if those effects extend to their pain ratings, nausea, and overall patient experience. Current research on use of steroids in rhinoplasty suggests that its use may decrease pain and nausea and benefit the patients overall experience.

Minimizing complications for any surgery is of upmost importance for surgeons.. However, the benefits of oral corticosteroid use for rhinoplasty patients in the immediate post-operative period are poorly understood and practice patterns vary widely. To identify and quantify the benefits and drawbacks of oral corticosteroid use in the immediate post-operative period for primary rhinoplasty patients, pain, swelling, nausea, patient experience, and post-operative swelling will be studied.

Rhinoplasty is a popular but challenging surgery. To date, there has been very little evidence on how using medrol in the postoperative period benefits a patient in terms of pain, nausea and their overall experience. The procedure is often associated with pain, edema, bruising and postoperative nausea. We currently do use oral corticosteroids for prevention of postoperative edema and ecchymosis however, we don't have a clear idea on how use of postoperative oral steroids effects pain, nausea and the overall patient experience. This study would like to add to the body of knowledge on oral corticosteroid use in the perioperative rhinoplasty period. It would be a simple, inexpensive study that may have significant benefit for future patients and surgeons. This medication is already used and has an established safety profile. This study would simply randomize patients to treatment vs placebo to determine if any real benefit exists, in an effort to determine if this practice should be standardized and universally applied in the future, or deemed unnecessary.

The prospective participants are patients who choose to undergo elective rhinoplasty surgery with one of three attending surgeons in the division of Facial Plastic Surgery within the Department of Otolaryngology/Head and Neck Surgery at Vanderbilt University Medical Center. Patients who elect to undergo surgery will be informed of the study and offered the opportunity to volunteer to participate in person either during the preoperative clinic visit OR in the preoperative area on the day of surgery. They will be led through an informed consent process, and excluded if they meet any of the exclusion criteria. Patients will be placed in the intervention group if their MRN is even and in the no intervention group if their MRN is odd.

The patients will be met on the day of surgery by a research coordinator, who is one of the study's KSP. The research coordinator will be responsible for screening the patients and determining eligibility based on the inclusion/exclusion criteria above. All participation will be strictly voluntary and will require informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age who elect to undergo cosmetic or functional open primary rhinoplasty with/without osteotomies (repositioning the nasal bones)
* No other facial plastics procedure nor sinus surgery performed simultaneously.

Exclusion Criteria:

* revision rhinoplasty
* diabetic patients
* patients with an allergy to steroids
* use of PPE implants
* parents receiving concurrent sinus surgery
* patients receiving biologics or preop oral steroids
* Patients that are pregnant or attempting to conceive
* Liver failure or cirrhosis
* Diagnosis of hypothyroidism
* Diagnosis of glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain level | Daily for 7 days
  Pain measured on a 5 point likert scale from no pain at all to worst pain ever experienced
Nausea | Daily for 7 days
  Nausea measured on 5 point likert scale from no pain at all to worst pain ever experienced
Edema | Daily for 7 days
  Edema measured based on a reference image. Edema rated based on how far from nose and eyes has any swelling dispersed.
Bruising | Daily for 7 days
  Bruising measured based on a reference image. Bruising rated based on how far from the nose and eyes did bruising extend to.

CONTACTS AND LOCATIONS:
Overall Officials: Priyesh N Patel, MD, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual patient data with other researchers.

REFERENCES:
- [Background] da Silva EM, Hochman B, Ferreira LM. Perioperative corticosteroids for preventing complications following facial plastic surgery. Cochrane Database Syst Rev. 2014 Jun 2;2014(6):CD009697. doi: 10.1002/14651858.CD009697.pub2. PMID 24887069
- [Background] Hwang SH, Lee JH, Kim BG, Kim SW, Kang JM. The efficacy of steroids for edema and ecchymosis after rhinoplasty: a meta-analysis. Laryngoscope. 2015 Jan;125(1):92-8. doi: 10.1002/lary.24883. Epub 2014 Aug 18. PMID 25131000
- [Background] Wu TJ, Huang YL, Kang YN, Chiu WK, Chen JH, Chen C. Comparing the efficacy of different steroids for rhinoplasty: A systematic review and network meta-analysis of randomized controlled trials. J Plast Reconstr Aesthet Surg. 2023 Sep;84:121-131. doi: 10.1016/j.bjps.2023.04.087. Epub 2023 May 3. PMID 37329745